CLINICAL TRIAL: NCT04794764
Title: Evaluation of Videolaryngoscopy (McGrath Mac) Compared to Direct Laryngoscopy for Rapid Sequence Intubation in Operating Room
Brief Title: Videolaryngoscopy Compared to Direct Laryngoscopy
Acronym: LARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Krankenhaus der Borromaerinnen Trier (Unknown); University Medical Center Freiburg (Other); BundeswehrZentralkrankenhaus Koblenz (Other); Krankenhaus Hetzelstift (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, PD Dr. med. habil. Marc Kriege, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JohannesGUV
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Aspiration of Gastric Contents
Keywords: Airway Management; Videolaryngoscopy; Adverse Events
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McGrath MAC (Experimental): First pass success rate using the McGrath Mac
  Interventions: Device: McGrath Mac
- Macintosh Laryngoscope (Experimental): First pass success rate using the Macintosh laryngoscope
  Interventions: Device: Macintosh Laryngoscope

INTERVENTIONS:
Device: McGrath Mac — in a randomized order we evaluate the first pass success rate of the tracheal tube into the trachea.
  Arms: McGrath MAC
Device: Macintosh Laryngoscope — in a randomized order we evaluate the first pass success rate of the tracheal tube into the trachea.
  Arms: Macintosh Laryngoscope

SUMMARY:
Videolaryngoscope (Macintosh-type blade) compared with direct laryngoscopy for rapid sequence intubation in the operating room

DETAILED DESCRIPTION:
Video laryngoscopy (VL) is a etablished method of achieving tracheal intubation and there is evidence to show that visualisation of larynx can be improved using VL in failed tracheal Intubation (NAP 4 Report). VL has been shown to improve first attempt success compared to direct laryngoscopy in many clinical settings including intensive care unit (ICU) and emergency department (ED). This is a proposed comparison study of a VL, use in patients with a high risk for pulmonary Aspiration and requiring tracheal Intubation. An national, multi-center, prospective randomized comparative trial is proposed testing the superiority of oral tracheal intubation with the McGrath® MAC versus conventional laryngoscope in adult patients under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years
* capacity to consent
* Present written informed consent of the research participant

Exclusion Criteria:

* Age <18 years
* Existing pregnancy
* Lack of consent
* inability to consent
* Difficult Airway / Defined Indications for awake intubation
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2021-07-24 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
First pass Intubation success rate | at intubation in 60 seconds
  successful tracheal intubation at the first attempt, compared to more than one attempt

SECONDARY OUTCOMES:
Time to ventilation | at intubation in 120 seconds
  From Insertion of the blase into the mouth until first ventilation
Cormack and Lehane Classification | < 120 seconds
  after insert the device the user describe the glottis visualisation
Overall success rate | < 120 seconds
  after two attempts using defined rescue techniques (e.g. rigid stylet, laryngeal mask)
Intubation difficult score | < 120 seconds
  Based on parameters known to be associated with difficult intubation (0=easy intubation to 5=difficult intubation
adverse events | after 24 hours
  sore throat
complications | < 120 seconds
  mucosal injury

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, PhD, Principal Investigator — University JG, Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Kriege M, Lang P, Lang C, Pirlich N, Griemert EV, Heid F, Wittenmeier E, Schmidtmann I, Schmidbauer W, Janig C, Jungbecker J, Kunitz O, Strate M, Schmutz A. Anaesthesia protocol evaluation of the videolaryngoscopy with the McGrath MAC and direct laryngoscopy for tracheal intubation in 1000 patients undergoing rapid sequence induction: the randomised multicentre LARA trial study protocol. BMJ Open. 2021 Oct 6;11(10):e052977. doi: 10.1136/bmjopen-2021-052977. PMID 34615684